CLINICAL TRIAL: NCT00512434
Title: Injection of Concentrated Autologous Bone-marrow (IMOCA) and Bone Union of Open Tibial Shaft Fracture: Randomized Study to Assess Efficiency of IMOCA in Addition to Standard of Care.
Brief Title: Percutaneous Autologous Bone-marrow Grafting for Open Tibial Shaft Fracture
Acronym: IMOCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRN/06/PR/IMOCA; ID RCB 2007 - A00032 - 51 (Other: AFSSAPS)
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Tibial Fractures; Fractures, Open
Keywords: tibial; shaft; fracture; open; bone-marrow; graft; injection; mesenchymal stem cell
MeSH Terms: conditions — Tibial Fractures; Fractures, Open; Fractures, Bone | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control in arm fields (Active Comparator): Standard treatment Intervention no'Osteosynthesis'
  Interventions: Procedure: Osteosynthesis
- IMOCA (Experimental): Intervention 'Osteosynthesis' Percutaneous autologous bone-marrow grafting - surgical technique (ref: Hernigou Ph et al J Bone Joint Surg Am ,2006; 88 (sup 1 part 2): 322-327
  Interventions: Procedure: Osteosynthesis

INTERVENTIONS:
Procedure: Osteosynthesis — Nail or external fixator Intervention 'Osteosynthesis'

SUMMARY:
The treatment of open tibial shaft fracture is often complicated by delayed union or non-union. The objective of this study is to evaluate the efficacy of autologous concentrated bone-marrow to accelerate healing of open tibial shaft fractures and to reduce the need for secondary intervention.

In a prospective, randomized, controlled, single-blind study, 186 patients with an open tibial will be randomized to receive either the standard of care (fixation by nail or external fixator and routine soft-tissue management), or the standard of care with percutaneous injection, one month after fracture, of autologous concentrated bone-marrow. Randomization will be stratified by severity of the open wound. The primary outcome measure will be the proportion of patients requiring secondary intervention because of delayed union or nonunion within twelve months post-fracture.

DETAILED DESCRIPTION:
This study will be conducted at 13 University Hospitals in France. The protocol has been approved by the institutional review board. After written informed consent, patients will be randomized, in the days after the fracture in 2 groups of 93 patients : 1) the control group (standard of care only: fixation by nail or external fixator and routine soft-tissue management) and 2) the study group (standard of care with percutaneous injection, one month after fracture, of autologous concentrated bone-marrow). Randomization will be stratified by severity of the open wound and by center. For the wound, strata A comprise Gustilo-Anderson types I, II and III-A and strata B, type III-B.

For the study group, the injection is scheduled at 1 month ± 5 days after the fracture. The techniques have been described by Hernigou (J Bone Joint Surg Am, 2006; 88(sup 1 part 2): 322-327). There are 3 steps: marrow aspiration (300 - 500 g) from iliac crest under general anesthesia, centrifugation in cell therapy unit to obtain a concentrated buffy coat of about 50 ml containing progenitor cells and other mononuclear cells, percutaneous injection in the fracture site of 20-30 ml of the buffy coat under fluoroscopy control.

Apart from the injection, the standard of care is the same for the 2 groups. Patients will be followed for 12 months, with assessments at 1, 2, 3, 6, 9 and 12 months.

All analysis will be based on the intent to treat the population. The primary outcome measure will be the proportion of patients requiring secondary intervention because of delayed union or nonunion within twelve months post fracture. An independent panel of surgeons will evaluate all secondary procedure with the potential of promoting fracture-healing.

An independent evaluation of fracture union will be conducted by a radiology panel blinded to treatment allocation and all other patient data.

An outcome will be considered to be successful when the fracture heal, according to the investigator, without secondary intervention and is radiographically united during patient follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 17 years or more
* Open tibial shaft fracture with Gustilo-Anderson type I, II, III A or B
* Written informed consent
* Affiliated to French Social Security

Exclusion Criteria:

* Circumferential bone loss
* Vascular or nerve injury
* Injury, other than tibial fracture, interfering with weight bearing
* Infection (skin, soft-tissue or bone)
* Disease or treatment interfering with bone union: head injury with coma, pathologic fracture
* Medical history on iliac wing contraindicating bone-marrow aspiration
* Corticoid or immunosuppressive therapy more than one week
* Pregnancy at the day of inclusion in study
* History of positive serology for HIV1+2, HBs, HCV
* Adult in the care of a guardian
* Impossibility to meet at the appointments for the follow-up

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-09; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients requiring secondary intervention because of delayed union or nonunion within twelve month post fracture. | one year

SECONDARY OUTCOMES:
Relation between the number of the progenitor available injected with concentrated bone marrow aspirated and the rate of bone union. | one year
Comparison of the rate of complications between the 2 groups. | one year
Economic impact study. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Rosset, Pr, Principal Investigator — Service d'orthopédie II - CHRU de Tours
Locations (11):
- France (11):
  - UH Angers, Angers
  - UH Besançon Jean Minjoz, Besançon
  - UH Brest Cavale Blanche, Brest
  - UH Clermont Ferrand Gabriel Montpied, Clermont-Ferrand
  - UH Grenoble Michallon Hospital, Grenoble
  - UH Grenoble South Hospital, Grenoble
  - UH Nancy Central Hospital, Nancy
  - UH Nantes Hôtel Dieu, Nantes
  - UH Pitié Salpétrière AH HP, Paris
  - UH Tours CHRU Trousseau, Tours
  - UHTOURS, Tours